CLINICAL TRIAL: NCT04411966
Title: Integrating 18F-FDG PET/CT With 18F-FLT PET/CT in Predicting Treatment Response and Prognosis of Metastatic/Recurrent Breast Cancer
Brief Title: Early Interim 18F-FDG-PET and 18F-FLT-PET for Predicting Treatment Response and Survival in Metastatic Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: CMRPG2C0483
Record Dates: First submitted 2020-05-12; First posted 2020-06-02 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2018-05

CONDITIONS: Metastatic Breast Cancer
Keywords: 18F-fluorothymidine; 18F-fluorodeoxyglucose; Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Participant received 18F-FLT and 18F-FDG at baseline, after 1st cycle , and after 2nd cycle of systemic chemotherapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 18F-fluorothymidine PET (Experimental): Patients receive fluorothymidine F-18 IV over 1 minute and undergo PET scan over 60 minutes at least 10 days prior to systemic chemotherapy, and at least 10 days after first and second cycles of systemic chemotherapy.
  Interventions: Diagnostic Test: 18F-fluorothymidine

INTERVENTIONS:
Diagnostic Test: 18F-fluorothymidine — Patients receive fluorothymidine F-18 IV over 1 minute and undergo PET scan over 60 minutes at least 10 days prior to systemic chemotherapy, and at least 10 days after first and second cycles of systemic chemotherapy.

SUMMARY:
We aim to investigate the value of 3'-deoxy-3'-18F-fluorothymidine (18F-FLT) and 18F-fluorodeoxyglucose (18F-FDG) positron emission tomography/computed tomography (PET/CT) for early prediction of treatment response and survival in patients with metastatic breast cancer after salvage therapy.

DETAILED DESCRIPTION:
Patients with metastatic breast cancer were enrolled and received PET/CT using 18F-FLT and 18F-FDG at baseline, after 1st cycle , and after 2nd cycle of systemic chemotherapy. The standard reference for treatment response was classified according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria for contrast-enhanced CT (CE-CT) after 3 months of systemic chemotherapy. The metabolic response on PET was assessed according to PET response criteria in solid tumors (PERCIST) criteria and was correlated to the treatment response, progression-free survival (PFS), and overall survival (OS).

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histological evidence of breast cancer of any stage
* Participants must be diagnosed with metastatic breast cancer
* Participants should be willing and able to have both PET-CT scans
* Participants should be eligible for and plan to undergo systemic chemotherapy and should be seen by a oncologist prior to beginning the study
* Participants should have the ability to understand and the willingness to sign a written informed consent document
* Participants must sign a study specific consent form prior to registration

Exclusion Criteria:

* Patients have been diagnosed with other malignancy
* Patients with uncontrolled intercurrent illness including, but not limited to, ongoing or active infection or significant inflammation at treatment site or psychiatric illness/social situations that would limit compliance with study requirements or whose lab values do not meet the criteria above are excluded
* Pregnant women are excluded from this study
* Breast feeding women are excluded from this study

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2017-08-30 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
Change in 18F-fluorothymidine (18F-FLT) and 18F-fluorodeoxyglucose (18F-FDG) maximal standardized uptake value (SUV) as response to therapy | Baseline, post 1-cycle and post 2-cycle (at least 10 days prior to or after systemic chemotherapy, each cycle is 28 days)
  The response to therapy would be determined by Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1) by contrast-enhanced computed tomography (CE-CT). The change of SUVmax between the responders and non responders on 18F-FLT and 18F-FDG would be compared.

SECONDARY OUTCOMES:
Compare Positron Emission Tomography Response Criteria in Solid Tumors (PERCIST) and European Organization for Research and Treatment of Cancer (EORCT) response by 18F-FLT-PET and 18F-FDG-PET for the prediction of anatomic treatment response | Baseline, post 1-cycle and post 2-cycle (at least 10 days prior to or after systemic chemotherapy, , each cycle is 28 days)
  We will use both EORTC and PERCIST criteria to compare the 18F-FLT-PET and 18F-FDG-PET metabolic response for the predictions of anatomic treatment response. Receiver operating characteristic (ROC) curve analysis and comparison were performed to evaluate the performance of 18F-FLT-PET and 18F-FDG-PET in predicting the anatomic treatment response, both with EORTC and PERCIST criteria.

OTHER OUTCOMES:
Progression-free survival (PFS) was defined as the time from the date of inclusion in the study to disease recurrence or progression. | Baseline, post 1-cycle and post 2-cycle (at least 10 days prior to or after systemic chemotherapy, each cycle is 28 days)
  Compare Positron Emission Tomography Response Criteria in Solid Tumors (PERCIST) and European Organization for Research and Treatment of Cancer (EORCT) response by 18F-FLT-PET and 18F-FDG-PET for the prediction of survival outcomes
Overall survival (OS) was defined as the time from the date of inclusion in the study to the date of death from any cause or last follow-up. | Baseline, post 1-cycle and post 2-cycle (at least 10 days prior to or after systemic chemotherapy, each cycle is 28 days)
  Compare Positron Emission Tomography Response Criteria in Solid Tumors (PERCIST) and European Organization for Research and Treatment of Cancer (EORCT) response by 18F-FLT-PET and 18F-FDG-PET for the prediction of survival outcomes

REFERENCES:
- [Derived] Su TP, Huang JS, Chang PH, Lui KW, Hsieh JC, Ng SH, Chan SC. Prospective comparison of early interim 18F-FDG-PET with 18F-FLT-PET for predicting treatment response and survival in metastatic breast cancer. BMC Cancer. 2021 Aug 10;21(1):908. doi: 10.1186/s12885-021-08649-z. PMID 34376155